CLINICAL TRIAL: NCT02243215
Title: Off-site vs. On-site Simulation Training in Laparoscopy a Randomized Trial
Brief Title: Off-site Training in Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: Region Capital Denmark (Other)
Responsible Party: Principal Investigator, Ebbe Thinggaard, Medical Doctor, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TABLT 2 Offsite; REG-68-2014 (Other: Regional Data Protection Agency)
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Off-site Training in Laparoscopy
Keywords: Laparoscopy; Training; Off-site; Box trainer; Virtual Reality Simulator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Offsite training (Experimental): Access to a portable trainer for laparoscopic skills
  Interventions: Other: Access to a portable trainer for laparoscopic skills
- Onsite training (No Intervention): Will be able practice on-site at Center of Clinical Education and at their local hospital.

INTERVENTIONS:
Other: Access to a portable trainer for laparoscopic skills — Participants will have a portable trainer available to allow training at their convenience, and will be able practice on-site at Center of Clinical Education and at their local hospital.
  Other Names: Laptap(R)
  Arms: Offsite training

SUMMARY:
The study is a randomized study exploring the difference between off-site vs. on-site training in laparoscopic skills. The study will be performed using fifty surgical trainees from the departments of urology, surgery and gynecology. The participants will be recruited, enrolled and randomized during the introductory course in basic laparoscopic techniques held six times annually at Center of Clinical Education(CEKU).

Participants will be able to train laparoscopic skills on a Box Trainer(BT) and on a Virtual Reality Simulator(VRS). They will practice until they reach a predefined level of proficiency on seven basic modules, the procedure module; "salpingectomy" on the LapSim™ and reach the passing level of 358pts on the Training and Assessment of Basic Laparoscopic Techniques(TABLT) technical test.

The intervention group will have a portable trainer available to allow training at their convenience, be it at home or at work. The control group will only practice on-site at CEKU and at their local hospital.

Participants will be asked to keep a training log with details of time spend on training and number of training sessions. The training log will contain information on any type practice involving laparoscopy be it on a BT or a VRS at the local hospital, at home on the tablet trainer or training at CEKU. Also time spend in the operation room, assisting or performing laparoscopic surgery will be registered.

To pass the TABLT all participants will book a test session at CEKU for their final test at the end of their training. At the test sessions TABLT test scores will be established on site by the Chief Investigator and afterwards using video recordings of the test. A blinded rater will give scores based on the video recordings and this will be the decisive rating to determine whether the participant has passed the test.

To pass the VRS training an employee at CEKU will monitor a VRS practice session in which proficiency level is reached.

The enrollment of participants is expected to finish June 2015 a data analysis will be performed in July 2015.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* hey have performed more than 50 laparoscopic procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Difference in time(days) to reach a defined proficiency level(358pts) on the TABLT technical test. | 6 months
Trainees use of off-site training in laparoscopic surgery | 6 months
  Qualitative focus group interviews, individual interviews and log-books

SECONDARY OUTCOMES:
Difference in time(mins.) used on training to reach a defined proficiency level(358pts) on the TABLT technical test. | 6 months
Difference in the number of training sessions used to reach a defined proficiency level(358pts) on the TABLT technical test. | 6 months
Difference in time(days) to reach a defined proficiency level on seven basic tasks and the salpingectomy module on the Lap Sim(R). | 6 months
Difference in time(mins.) used on training to reach a defined proficiency level on seven basic tasks and the salpingectomy module on the Lap Sim(R). | 6 months
Difference in number of training sessions used to reach a defined proficiency level on seven basic tasks and the salpingectomy module on the Lap Sim(R). | 6 months
Correlation between participants rating of pre-tests and a blinded rater | 6 months

OTHER OUTCOMES:
Difference in number of laparoscopic surgeries in 6 month period after having passed the TABLT test and reached a defined proficiency level on seven basic tasks and the salpingectomy module on the Lap Sim(R). | 6 months
Difference in test score on the TABLT technical test. | 6 months
Difference in number of laparoscopic surgeries during the training period, from enrollment to having passed the TABLT test | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ebbe Thinggaard, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Center for Clinical Education, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Background] Korndorffer JR Jr, Bellows CF, Tekian A, Harris IB, Downing SM. Effective home laparoscopic simulation training: a preliminary evaluation of an improved training paradigm. Am J Surg. 2012 Jan;203(1):1-7. doi: 10.1016/j.amjsurg.2011.07.001. PMID 22172481
- [Background] Ericsson KA. Deliberate practice and the acquisition and maintenance of expert performance in medicine and related domains. Acad Med. 2004 Oct;79(10 Suppl):S70-81. doi: 10.1097/00001888-200410001-00022. No abstract available. PMID 15383395
- [Background] Gallagher AG, Jordan-Black JA, O'Sullivan GC. Prospective, randomized assessment of the acquisition, maintenance, and loss of laparoscopic skills. Ann Surg. 2012 Aug;256(2):387-93. doi: 10.1097/SLA.0b013e318251f3d2. PMID 22580935
- [Background] Strandbygaard J, Bjerrum F, Maagaard M, Winkel P, Larsen CR, Ringsted C, Gluud C, Grantcharov T, Ottesen B, Sorensen JL. Instructor feedback versus no instructor feedback on performance in a laparoscopic virtual reality simulator: a randomized trial. Ann Surg. 2013 May;257(5):839-44. doi: 10.1097/SLA.0b013e31827eee6e. PMID 23295321
- [Background] Snyder CW, Vandromme MJ, Tyra SL, Hawn MT. Proficiency-based laparoscopic and endoscopic training with virtual reality simulators: a comparison of proctored and independent approaches. J Surg Educ. 2009 Jul-Aug;66(4):201-7. doi: 10.1016/j.jsurg.2009.07.007. PMID 19896624
- [Background] Kahol K, Leyba MJ, Deka M, Deka V, Mayes S, Smith M, Ferrara JJ, Panchanathan S. Effect of fatigue on psychomotor and cognitive skills. Am J Surg. 2008 Feb;195(2):195-204. doi: 10.1016/j.amjsurg.2007.10.004. PMID 18194679
- [Derived] Thinggaard E, Bjerrum F, Strandbygaard J, Konge L, Gogenur I. A randomised clinical trial of take-home laparoscopic training. Dan Med J. 2019 Jan;66(1):A5525. PMID 30573006